CLINICAL TRIAL: NCT02058680
Title: A Phase 1A/1B, Two-Stage Study of a PSA/IL-2/GM-CSF Vaccine for the Treatment of PSA Recurrent Prostate Cancer in Hormone-Naive and Hormone-Independent Patients
Brief Title: Phase 1A/1B Study of PSA/IL-2/GM-CSF Vaccine for Recurrent Prostate Cancer in Hormone Naive and Hormone Independent Patients
Acronym: PSA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: OncBioMune Pharmaceuticals (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O11-10678; Department of Defense (Other Grant/Funding Number: DOD W911QY-11-C-0102)
Record Dates: First submitted 2014-02-04; First posted 2014-02-10 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer
Keywords: prostate specific antigen (PSA)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PSA/IL-2/GM-CSF vaccine (Experimental): In Stage 1 (Phase 1A), patients receive intradermal injections of PSA/IL-2/GM-CSF vaccine at Weeks 1, 2, 3, 7, 11, and 15.
  In Stage 2 (Phase 1B), patients will receive the same course of vaccine (induction as in Phase 1A; this will be followed in eligible patients by maintenance vaccinations alternating between IL-2 alone at Weeks 23, 31, and 39) and complete vaccine (PSA/IL-2/GM-CSF) at Weeks 27, 35, and 43.
  Interventions: Biological: PSA/IL-2/GM-CSF

INTERVENTIONS:
Biological: PSA/IL-2/GM-CSF — In Stage 1 (Phase 1A), patients receive intradermal injections of PSA/IL-2/GM-CSF vaccine at Weeks 1, 2, 3, 7, 11, and 15.
  In Stage 2 (Phase 1B), patients will receive the same course of vaccine (induction as in Phase 1A; this will be followed in eligible patients by maintenance vaccinations alternating between IL-2 alone at Weeks 23, 31, and 39) and complete vaccine (PSA/IL-2/GM-CSF) at Weeks 27, 35, and 43.

SUMMARY:
This study is investigating the safety and efficacy of a vaccine directed against prostate tumor cells. The researchers are interested in evaluating the safety and tolerability of the vaccine, and the effects of the vaccine on survivability, time to measurable disease, prostate-specific antigen (PSA) level in the blood, and the immune response to the vaccine.

Eligible patients include those with recurrent prostate cancer as shown by elevated levels of PSA, although there is no evidence of tumors that are measurable by imaging studies. In addition, to be eligible patients must have prostate cancer that either has not been treated by hormonal therapy or is not responsive to hormonal therapy.

DETAILED DESCRIPTION:
In Phase 1A, hormone naive and hormone independent patients are enrolled in a 1:1 ratio. All patients receive intradermal injections of the PSA/IL-2/GM-CSF induction vaccine at Weeks 1, 2, 3, 7, 11 and 15.

In Phase 1B, which will be initiated after Phase 1A, will first receive the induction vaccine (PSA/IL-2/GM-CSF) according to the same schedule as patients in Phase 1A. Then, in eligible Phase 1B patients, following the induction vaccine regimen, alternating maintenance vaccination will be administered as follows: at Weeks 23, 31, and 39, IL-2 alone will be administered; at Weeks 27, 35, and 43, the complete vaccine (PSA/IL-2/GM-CSF) will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Age greater than18 years
* Rising serum PSA levels documented by 3 values over the last 6 months prior to study enrollment. Each value must be greater than 2 weeks from the previous value.
* Patients with rising PSA must have had either 1) prior definitive therapy including surgery or radiation therapy (hormone-naïve, defined as hormone-naïve patients and patients who received hormone therapy in the past who currently have total testosterone greater than 50 ng/dL), or 2) hormone suppressive therapy as documented by surgical castration or a serum testosterone value less than 50 ng/dL (hormone-independent). Patients must have completed these therapies for at least 6 months but no longer than 20 years prior to enrollment
* PSA value within 4 weeks of starting therapy less than 20 ng/mL for hormone-naïve patients (defined as hormone-naïve patients and patients who received hormone therapy in the past who currently have total testosterone greater than 50 ng/dL) or less than 60 ng/mL for hormone-independent patients.
* Patients must have the following laboratory values: ANC greater than 1500/mcL, platelet count greater than 100,000/mcL, hemoglobin greater than 10 g/dL, bilirubin less than 1.5 x upper limits of normal, AST less than 1.5 x upper limits of normal
* Patients must have adequate lung function, as defined by oxygen saturation greater than or equal to 90% by pulse oximetry
* Patients must have QTc interval less than 450 msec
* Patients must have adequate EGFR greater than 30 mL/min per 1.73 m2 (per VA formula and adjusted for gender and race)
* Patients with female partners of childbearing potential must use at least one form of Investigator-approved contraception while on-study and for 30 days after their last administration of study investigational therapy. Acceptable birth control options include: a) surgical sterilization (subject and/or subject's partner), b) approved hormonal contraceptives or therapies (such as birth control pills, Depo-Provera, or Lupron Depot), c) barrier methods (such as a condom or diaphragm) used with a spermicide, and d) an intrauterine device (IUD).

Exclusion Criteria:

* Presence of documented neuroendocrine differentiation on the original pathology report
* Evidence of metastatic disease
* Immune compromised patients including but not limited to: systemic immune suppressive medications within 6 weeks of enrolling; HIV-positive and below normal CD4 lymphocytes (less than 500 cells per microliter). Patients must be tested for HIV seropositivity and CD4 lymphocyte count to be eligible for the study
* Prior malignancy. Patients with nonmelanoma skin cancer or other cancers with greater than 3 years without evidence of disease recurrence are eligible
* Inability to give informed consent
* Any condition that, according to the investigator, would make the patient an inappropriate study candidate.
* Patients with pulmonary disease limiting daily function or requiring oxygen supplementation
* Patients with significant cardiac disease including heart failure that meets New York Heart Association (NYHA) class III and IV definitions, history of myocardial infarction within six months of study entry, uncontrolled dysrhythmias, or QTc greater than or equal to 450 msec
* Patients with existing autoimmune disorders (IL-2 and GM-CSF carry a theoretical clinical risk of exacerbating underlying autoimmune disorders)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Adverse Events | From first injection until 30 days past the last injection

SECONDARY OUTCOMES:
PSA Doubling Time (PSADT) and PAP levels | Measured at pretreatment screening, prior to first vaccine injection, and then following vaccination at treatment Weeks 7, 15, 19 (Phase 1A), and then every 12 weeks up to Week 103 (Phase 1B).
Time to measurable disease | Time to confirmation of disease recurrence. Patients undergo bone scans and CT scans of chest, abdomen, and pelvis at pretreatment and then at Week 19, and every 24 weeks (6 months) until Week 105.
Time to subsequent therapy | Time (days) from Day 1 (first day of vaccine treatment) to either the next investigational anticancer treatment or the first supplemental palliative treatment, up to Week 105.
Overall survival | Time (days) from Day 1 to the patient's death. Patients will be followed up to Week 105.
Vaccine-induced immune response including antiPSA antibodies, lymphocyte activation assays, and serum and intracellular cytokine levels | Measured at pretreatment screening or Day 1 pre-vaccination, and then treatment Weeks 7 and 19, and then every 12 weeks up to Week 103

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Wang-Rodriguez, MD, Principal Investigator — University of California, San Diego; Gregory A Daniels, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States